CLINICAL TRIAL: NCT06752499
Title: Individualized rTMS Concurrent With Motor Actions Promotes Post-stroke Upper Limb Recovery
Brief Title: rTMS Combined With Motor Training for the Treatment of Upper Limb Motor Dysfunction in Stroke Patients
Acronym: rTMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Changhai Hospital (Other); Shanghai Yangzhi Rehabilitation Hospital (Unknown); shanghai center for brain science and brain-inspired technology (Unknown)
Responsible Party: Principal Investigator, Qing Xie, PhD, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022361
Record Dates: First submitted 2024-12-27; First posted 2024-12-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Upper Extremity Paresis
Keywords: Repetitive Transcranial Magnetic Stimulation; Upper Limb Motor Dysfunction; online; motor task training; individualized; Motor evoked potentials
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online stimulation (Experimental): 5 Hz rTMS is applied to the primary motor cortex on the affected hemisphere when the patients are performing motor tasks.
  Interventions: Device: Online stimulation
- Offline stimulation (Active Comparator): After 5 Hz rTMS is applied to the primary motor cortex on the affected hemisphere, the patients perform motor tasks.
  Interventions: Device: Offline stimulation
- Sham stimulation (Sham Comparator): Sham rTMS is applied to the primary motor cortex on the affected hemisphere when the patients are performing motor tasks.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Online stimulation — 5 Hz rTMS is applied to the primary motor cortex on the affected hemisphere when the patients are performing motor tasks.
  Arms: Online stimulation
Device: Offline stimulation — After 5 Hz rTMS is applied to the primary motor cortex on the affected hemisphere, the patients perform motor tasks.
  Arms: Offline stimulation
Device: Sham stimulation — Sham rTMS is applied to the primary motor cortex on the affected hemisphere when the patients are performing motor tasks.
  Arms: Sham stimulation

SUMMARY:
The goal of this clinical trials is to investigate the effectiveness of online repetitive transcranial magnetic stimulation (rTMS) in enhancing upper limb motor rehabilitation during the subacute and chronic phase of stroke. It will also learn about the safety of online rTMS intervention methods. The main questions it aims to answer are:

1. Does rTMS combined with motor training improve motor rehabilitation in patients？
2. Does repetitive transcranial magnetic stimulation (rTMS) combined with motor training enhance the upper limb motor rehabilitation ability in stroke patients by strengthening the functional coupling of the motor circuit to achieve functional reorganization of the brain network ?

Researchers will compare online rTMS to offline and sham stimulation in stroke patients to see if online rTMS works to alleviate motor dysfunction in multicenter multicenter, blinded and controlled trial.

Participants will:

1. randomized to one group(online, offline or sham);
2. receive rTMS treatment for 10 days, with 5 working days per week for a total of two weeks;
3. receive magnetic resonance imaging (MRI) and electroencephalogram (EEG) evaluations before and after the entire treatment;
4. conduct scales and MEP assessment one day before the treatment, as well as one day, one month, and three months after the treatment.

DETAILED DESCRIPTION:
In this study, patients were be randomly assigned to three groups: online, offline and sham groups. if patients were able to induce MEPs, intensity of TMS will be 80% RMT; if not , inensity of TMS will be 70%~80% of TMS output.

Patients were stimulated over 2 week period, 4 sessions of tasks were performed everyday. The patient will undergo a 2-week (10-day) stimulation protocol, with fourty tasks performed daily. This includes one session of 10 baseline tasks measurement and three sessions of 5 Hz rTMS synchronized with 10 motor tasks. rTMS will be applied to the ipsilesional motor cortex.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is first diagnosed with stroke through neurological examination, CT or MRI scan.
2. The vital signs are stable and there is a certain degree of upper limb motor dysfunction.
3. The age is between 20 and 80 years old.
4. The cognitive ability is not significantly affected and the patient can cooperate with various examinations and assessments, with a MMSE score ≥ 20 points.
5. There are no serious complications (such as pneumonia, heart failure, urinary tract infection or malnutrition).
6. There is no pathological condition that is a contraindication for TMS in the medical history (for example, patients with metal in the brain, such as aneurysm clips, patients with a cardiac pacemaker, pregnant women, or those with a history of epileptic seizures).
7. The patient or guardian agrees to sign the informed consent form.

Exclusion Criteria:

1. Patients with severe heart, lung, liver, kidney diseases and malignant tumors;
2. Those with a history of aphasia, severe cognitive impairment or mental illness;
3. Patients who have had a history of epileptic seizures in the last month or are taking anti-epileptic drugs recently;
4. Those with severe visual or hearing impairments, unable to communicate normally;
5. People with metal implants, pacemakers, skull defects or other conditions that prevent them from undergoing TMS.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean Change in FM-UE From Baseline | Day 105 （three months after 2-week intervention）
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment.
  The Fugl-Meyer Assessment - Upper Extremity (FMA-UE) is the upper limb motor domain includes items assessing movement, coordination, and reflex action of the shoulder, elbow, forearm, wrist, hand. It ranges from 0 (hemiplegia) to 66 points (normal motor performance).
  FM-UE scale was assessed by site raters who were masked to the intervention).

SECONDARY OUTCOMES:
Mean Change in ARAT score from Baseline | Day 105 （three months after 2-week intervention）
  The Action Research Arm Test (ARAT) is a 19 item observational measure used by physical therapists and other health care professionals to assess upper extremity performance (coordination, dexterity and functioning) in stroke recovery, brain injury and multiple sclerosis populations. The ARAT was originally described by Lyle in 1981 as a modified version of the Upper Extremity Function Test and was used to examine upper limb functional recovery post damage to the cortex.
  ARAT score was assessed by site raters who were masked to the intervention.
Mean Change in WMFT score from Baseline | Day 105 （three months after 2-week intervention）
  The WMFT is used to assess the upper limb motor function of patients and serves as an effective supplement to the FMA-UE. By timing single-joint movements, multi-joint movements, and functional activities, as well as evaluating movement quality and speed, it can quantitatively assess the upper limb motor ability of stroke patients. It is more sensitive to patients with mild to moderate stroke, and its grading is relatively detailed, which can sensitively reflect the subtle changes in patients' motor function during evaluation.
  The WMFT consists of 15 items, among which items 1-6 are simple joint movements, and items 7-15 are complex functional actions. This scale can not only evaluate impairments but also assess the effect of training on disabilities. The WMFT has good validity and reliability and can be used to evaluate the upper limb function of stroke patients.
  WMFT score was assessed by site raters who were masked to the intervention.
Mean Change in MBI score from Baseline | Day 105 （three months after 2-week intervention）
  The Barthel Index for activities of daily living was introduced in 1965 by Barthel and Mahoney to be used in the assessment of the degree of assistance required by patients with stroke (other neuromuscular or musculoskeletal disorders or oncology patients) with regards to 10 items of mobility and self-care (ADL).
  MBI score was assessed by site raters who were masked to the intervention.
Mean Change in PSQI score from Baseline | Day 105 （three months after 2-week intervention）
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval.
  The PSQI is commonly used in both clinical and research settings to evaluate various aspects of sleep. It is a valuable tool for assessing sleep quality as it captures multiple dimensions of sleep, including both subjective experiences and objective parameters. It allows researchers and healthcare providers alike to obtain a comprehensive understanding of an individual's sleep patterns and disturbances and inform treatment decisions and interventions for sleep disorders.
  PSQI score was assessed by site raters who were masked to the intervention).
Motor Evoked Potential (MEP) - Resting Motor Threshold (RMT) | Before intervention (Week 0); In the middle of intervention (Week 1); After intervention (Week 2); Follow-up 1 (one month after intervetnion); Follow-up 2 (three months after intervention)
  Resting motor threshold is an objective measure of cortical excitability. Numerous studies indicate that the success of motor recovery after stroke is significantly determined by the direction and extent of cortical excitability changes.
The average completion time for baseline tasks | Before intervention (Week 0); Middle of intervention (Week 1); After intervention (Week 2)
  The average completion time for baseline tasks refers to the time (seconds) taken by the patient to complete the baseline motor task before each intervention.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shanghai Ruijin Hospital, affiliated to Shanghai Jiao Tong University, School of medicine, Shanghai, Shanghai Municipality
  - Shanghai Yang Zhi Rehabilitation Hospital, Shanghai, Songjiang
  - Changhai Hospital, Shanghai, Yangpu

IPD SHARING:
Plan to Share IPD: Yes
This study plans to share individual participant data with qualified researchers under specific conditions. Please refer to https://zenodo.org/records/17345584
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Authorized professional researchers, including but not limited to researchers engaged in neuroscience research who have obtained data access permission from their affiliated institutions, and clinical doctors from other medical institutions that have a cooperative relationship with this study and have signed data confidentiality agreements.
  They can access the detailed clinical medical histories of the participants, including past disease histories and treatment process records; neurological function assessment scale data; as well as imaging data collected during the study, such as brain magnetic resonance imaging (MRI) results. However, sensitive information related to participants' privacy, such as names, ID numbers, and contact information, will be strictly anonymized to ensure that such information cannot be obtained.
  They can contact the corresponding author or the first author via email.
URL: https://zenodo.org/records/17345584